CLINICAL TRIAL: NCT05488522
Title: A Phase I Study of SBRT Vaccination With Atezolizumab and Bevacizumab for Patients With Advanced Hepatocellular Carcinoma
Brief Title: SBRT With Atezo/Bev for HCC
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 851667; 851667 (Other: IRB)
Record Dates: First submitted 2022-07-19; First posted 2022-08-04 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Radiosurgery; atezolizumab; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- study treatment plan (Experimental): Patients will be enrolled in a Rolling 6 clinical trial design1. This study design retains sensitivity to identifying DLTs while having the benefit of decreasing accrual time given the long DLT period required to assess radiation toxicity. In this trial design, up to 6 patients can be enrolled at a time onto a dose level while awaiting DLT assessment. Established rules guide the decision for enrolling onto the current, next highest, or previous dose level based on the number of participants currently enrolled in a given cohort, the number of radiation-attributable dose-limiting toxicities (ra-DLTs) observed, and the number of patients with immature toxicity data. If the MTD is not reached after 6 patients have enrolled on dose level 3 (three 17Gy fractions of SBRT) and have completed toxicity evaluations, then the recommended phase 2 dose will be determined based on an analysis of the efficacy of the combination
  Interventions: Biological: SBRT + atezolizumab and bevacizumab

INTERVENTIONS:
Biological: SBRT + atezolizumab and bevacizumab — Stereotactic Body Radiotherapy (SBRT) is a radiation procedure that delivers precise doses of radiation in fractions. See following section for more information on the schedule, dose, volume, and simulation of SBRT.
  Atezolizumab is an FDA-approved immune checkpoint inhibitor that is used in the treatment of advanced HCC. It is administered as a flat-dose 1200 mg intravenous infusion every three weeks.
  Bevacizumab is an FDA-approved anti-VEGF monoclonal antibody that is used in the treatment of advanced HCC in combination with atezolizumab. It is administered as a weight-based dose of 15 mg/kg intravenous infusion every 3 weeks.

SUMMARY:
A phase I dose escalation and pharmacodynamic study of repeated dose stereotactic body radiotherapy (SBRT) administered with concurrent atezolizumab and bevacizumab for patients with advanced hepatocellular carcinoma (HCC)

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have hepatocellular carcinoma (HCC) that is not amenable to curative-intent surgical or ablation (where surgery or ablation are not indicated due to disease extent, co-morbidities, or other technical reasons) and systemic therapy is indicated.

Exclusion Criteria:

-

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Primary Objective | 3 years
  we will measure the total number of subjects that can tolerate the recommended phase II regimen of SBRT with atezolizumab/bevacizumab (atezo/bev) in patients with advanced hepatocellular carcinoma and the proportion of patients experiencing a radiation-attributable DLT at each dose level.

SECONDARY OUTCOMES:
Secondary Objective | 3 years
  To assess efficacy and safety, in terms of tumor objective response rate (ORR) by RECIST 1.1 and iRECIST
Overall Survival | 5 years
  we will be measuring for Overall Survival (OS) post study treatment.
Progression Free survival | 5 years
  We will be measuring for progression free survival with RECIST 1.1 definition

CONTACTS AND LOCATIONS:
Overall Officials: Edgar Ben-Josef, MD, Principal Investigator — Abramson Cancer Center
Locations (1):
- Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No